CLINICAL TRIAL: NCT04374331
Title: The Effect of Video-Assisted Training on Upper Extremity Problems and Functions in Patients Undergoing Rotator Cuff Repair: A Randomized Controlled Trial
Brief Title: Effect of Video-Assisted Training on Upper Extremity Problems and Functions in Patients Undergoing Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Gulay ALTUN UGRAS, Associate professor, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Gulay Altun
Record Dates: First submitted 2020-04-29; First posted 2020-05-05 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Rotator Cuff Repair
Keywords: Rotator cuff repair; video-assisted training; upper extremity problems; upper extremity functions; complication
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: prospective, parallel, two arm, randomized controlled clinical trial
Who Masked: Participant
Masking Description: Before inclusion, the patients were informed about the duration of care as usual, which could be six weeks or three months. The patients were blinded to the group assignment due to the nature of the intervention. The researchers involved in the data analysis and statistics stages were blinded to the group assignment, too. However, those involved in the running of the study were not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-Assisted Training Group (Experimental): The patients in the VAT group watch a training video in the patient rooms before RCR in addition to the routine treatment and care in the unit.
  Interventions: Other: video-assisted training
- control group (No Intervention): The control group received the routine treatment and care in the unit. The routine treatment and care of the unit includes verbal briefing by physicians and nurses about the surgical procedure before RCR, cold application and analgesic application for pain control after RCR, using arm sling, verbal discharge training (e.g., drug use, exercises, follow-up time, etc.) and discharge on the first post-operative day in the absence of complications. In addition, patients are invited to weekly controls to explain how to do the exercises and, if necessary, they are referred to physiotherapy.

INTERVENTIONS:
Other: video-assisted training — The patients in the VAT group watch a training video in the patient rooms before RCR. The VAT prepared by the researchers consisted of information about things to pay attention to in the hospital in the early period after RCR (nursing care on post-operative day 1, early mobilization, pain control, shoulder protection, and wearing/removing the shoulder sling), maintaining ADL at home (bathing, nutrition, eating, sleeping position, driving, doing household chores, sexual life, worship, and safety measures to be taken at home) and gradual exercise programs (for the first 90 days after discharge).
  Other Names: Control group
  Arms: Video-Assisted Training Group

SUMMARY:
This randomized controlled trial evaluates the effect of video-assisted training (VAT) on upper extremity problems and functions in rotator cuff repair (RCR) patients. The hypothesis of this study is that VAT decreases upper extremity problems and increases functions after RCR.

DETAILED DESCRIPTION:
Methods: Forty-eight elective RCR patients were randomly assigned to VAT and control groups. VAT group (n=24) received VAT including early post-operative care for RCR, activities of daily living (ADL) and gradual exercise program while control group (n=24) received routine care. Primary outcomes were upper extremity problems and functions, assessed using Disabilities of the Arm, Shoulder and Hand (DASH) and Modified Constant-Murley (MCM) scores. Secondary outcomes were complications within three months. Outcomes were collected at baseline, after six weeks and three months.

ELIGIBILITY:
Inclusion Criteria: Patients who

* underwent elective RCR for the first time;
* whose arm was suspended and fixed for up to three weeks after RCR;
* had an SMMT score of ≥23 points;

Exclusion Criteria: Patients who

* had been diagnosed with a psychiatric illness;
* have any history of an upper extremity fracture or a rheumatologic disease;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
Change upper extremity problems | Change from baseline the Disabilities of the Arm, Shoulder and Hand score at 3 months
  The patients' upper extremity problems were assessed using the Disabilities of the Arm, Shoulder and Hand. The possible scores on each part of the questionnaire range from 0 to 100, with higher scores indicating a higher disability level of patients (0=no disability, 100=maximum disability)
Change upper extremity functions | Change from baseline the Modified Constant-Murley score at 3 months
  The patients' upper extremity functions were assessed using the Modified Constant-Murley score. The Modified Constant-Murley score consists of 100 points in total: 15 points for pain, 20 points for daily of living activities, 40 points for movement and 25 points for strength. The maximum MCM score is 100 points, with higher scores indicating better shoulder functions

SECONDARY OUTCOMES:
Change of complications | 1st and 3rd months
  Determine complications after rotator cuff repair

CONTACTS AND LOCATIONS:
Overall Officials: Gulay Altun Ugras, PhD, Study Director — Mersin University
Locations (1):
- Mersin University, Mersin, Yenisehir, Turkey (Türkiye)